CLINICAL TRIAL: NCT01898143
Title: Cardiorespiratory Response During Whole Body Vibration Training in Patients With Chronic Obstructive Pulmonary Disease (COPD) or Interstitial Lung Disease (ILD)
Brief Title: Cardiorespiratory Response During Whole Body Vibration Training in Patients With Chronic Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head Physican (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: SpiroErgoGalileo-2013
Record Dates: First submitted 2013-06-24; First posted 2013-07-12 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Lung Disease (n=10); Interstitial Lung Disease (n=10)
Keywords: Whole body vibration, cardiorespiratory response
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole body vibration in COPD (Other): Patients with COPD GOLD III or IV
  Interventions: Other: Whole body vibration
- Whole body vibration in ILD (Other): PAtients with interstitial lung disease
  Interventions: Other: Whole body vibration

INTERVENTIONS:
Other: Whole body vibration

SUMMARY:
Whole body vibration training seems to be a useful adjunct in exercise training in patients with severe COPD. The basic principle relies on reflectory muscle contractions caused by a vibration stimulus. Until now the impact of whole body vibration training on cardiopulmonary parameters remained unknown. Therefore aim of this study is to investigate cardiopulmonary parameters during whole body vibration training in patients with chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

* COPD stage III or IV according to the Global Initiative for chronic obstructive lung disease [GOLD])
* Interstitial Lung disease (forced vital capacity (FVC) < 70% pred., diffusion capacity of lung for carbon monoxide (DLCO) 30-70% pred.)

Exclusion Criteria:

* Oxygen therapy during exercise required
* Severe exacerbation of lung disease, with necessity of change in medication or persistent symptoms > 3days
* activated arthrosis /arthropathy/ rheumatoid Arthritis/ acute discopathy
* acute thrombosis
* acute musculoskeletal inflammation
* Epilepsy
* Gallstones

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
peak oxygen consumption (VO2 peak) | during 1 exercise session
  subjects perform several short bouts (1 to 3 minutes duration) of squatting exercise with or without whole body vibration. The peak values of each single part is used for comparison.

SECONDARY OUTCOMES:
heart rate (HR) | during 1 exercise session
  subjects perform several short bouts (1 to 3 minutes duration) of squatting exercise with or without whole body vibration. The peak values of each single part is used for comparison.
minute ventilation (VE) | during 1 exercise session
  subjects perform several short bouts (1 to 3 minutes duration) of squatting exercise with or without whole body vibration. The peak values of each single part is used for comparison.
perceived exertion for dyspnea and leg fatigue (Borg-scale) | during 1 exercise session
  subjects perform several short bouts (1 to 3 minutes duration) of squatting exercise with or without whole body vibration. The peak values of each single part is used for comparison.
Alveolar-arterial oxygen difference (AaDO2) | during 1 exercise session
  subjects perform several short bouts (1 to 3 minutes duration) of squatting exercise with or without whole body vibration. The peak values of each single part is used for comparison.
breathing frequency (BF) | during 1 exercise session
  subjects perform several short bouts (1 to 3 minutes duration) of squatting exercise with or without whole body vibration. The peak values of each single part is used for comparison.
peak carbon-dioxide consumption (VCO2 peak) | during 1 exercise session
  subjects perform several short bouts (1 to 3 minutes duration) of squatting exercise with or without whole body vibration. The peak values of each single part is used for comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany